CLINICAL TRIAL: NCT04510259
Title: Selective Trunk Brachial Plexus Block: A Prospective Non-Randomized Study Intervention
Brief Title: Selective Trunk Brachial Plexus Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof Manoj K Karmakar, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SeTB
Record Dates: First submitted 2020-08-07; First posted 2020-08-12 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Upper Extremity Problem
Keywords: Brachial Plexus Block; Upper extremity
MeSH Terms: interventions — Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Selective Brachial plexus block (Experimental): Selective brachial plexus block will be done under ultrasound guidance to patients scheduled for upper extremity surgeries. Local anesthetic agents (a mixture of 2% lidocaine with 1:200,000 epinephrine and 0.5% levobupivacaine in a total of 25ml) will be injected at the superior, middle, and inferior trunks of the brachial plexus in order to anesthesize the whole upper limb.
  Interventions: Procedure: Selective Brachial plexus Block

INTERVENTIONS:
Procedure: Selective Brachial plexus Block — It is one type of peripheral nerve blocks for upper extremity surgery. In this study, the block will be done under the ultrasound guidance and the local anesthetic agent (a mixture of 2% Xylocaine with 1: 200,000 adrenaline and 0.5% Chirocaine in a total of 25ml) will be injected at the trunks of the brachial plexus in order to produce the surgical anesthesia of the whole upper extremity of the patients scheduled for upper limb surgeries.
  Other Names: Drug

SUMMARY:
Brachial plexus block (BPB) is frequently used as the sole anesthestic technique for upper extremity surgery. However, the choice of injection can be made from different approaches that often depends on the site of surgery because the extent of sensory-motor blockade after a BPB varies with the approach used. The investigator is not aware of any single BPB technique that can consistently produce surgical anaesthesia of the whole ipsilateral upper extremity. However, occasionally surgery entails that the whole upper extremity is anesthetized, i.e. from the shoulder to the elbow, or even the forearm, wrist or hands. This clinical challenge has been addressed previously using a combination of BPB techniques. The investigator has recently demonstrated that it is feasible to accurately identify majority of the main components of the brachial plexus above the clavicle, including the three trunks, using ultrasound imaging. Since majority of the innervation of the upper extremity, i.e. shoulder, arm, elbow, forearm, wrist and hand, originates from the three trunks of the brachial plexus, the investigator hypothesized that selectively blocking upper, middle, and inferior trunks of the brachial plexus will produce surgical anesthetsia of the whole ipsilateral upper extremity. The aim of this study is to assess a novel brachial plexus block technique, the selective trunk block (SeTB), and provide preliminary clinical evidence of its effectiveness in producing surgical anesthesia of the whole ipsilateral upper extremity.

DETAILED DESCRIPTION:
Brachial plexus block (BPB) is frequently used as the sole anesthetic technique for upper extremity surgery. The choice of technique often depends on the site of surgery because the extent of sensory-motor blockade after a BPB varies with the technique used. The investigator is not aware of any single BPB technique that can consistently produce surgical anesthesia of the whole ipsilateral upper extremity. However, occasionally surgery entails that the whole upper extremity is anesthetized, i.e. from the shoulder to the elbow, or even the forearm, wrist or hands. This clinical challenge has been addressed previously using a combination of BPB techniques. The investigator has recently demonstrated that it is feasible to accurately identify majority of the main components of the brachial plexus above the clavicle, including the three trunks, using ultrasound imaging. Since majority of the innervation of the upper extremity, i.e. shoulder, arm, elbow, forearm, wrist and hand, originates from the three trunks of the brachial plexus, the investigator hypothesized that selectively blocking upper, middle and inferior trunks of the brachial plexus will produce surgical anesthesia of the whole ipsilateral upper extremity, except for the area innervated by the intercostobrachial nerve (T2- medial aspect of the upper arm). In addition, there may be a potential advantage that phrenic nerve can be spared, so this blockade will not affect the respiratory function as it is common to see phrenic nerve palsy after interascalene BPB (100%) and supraclavicular BPB (50-67%). The aim of this study is therefore to assess a novel brachial plexus block technique, the "selective trunk block" (SeTB), and provide preliminary clinical evidence of its effectiveness in producing surgical anesthesia of the whole ipsilateral upper extremity.

ELIGIBILITY:
Inclusion Criteria:

* Elective upper extremity surgery
* Emergency upper extremity surgery

Exclusion Criteria:

* Patient refusal
* Local skin site infection
* Allergy to local anaesthetics
* Peripheral neuropathy
* Brachial plexopathy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2021-07-27 (Actual)

PRIMARY OUTCOMES:
Changes of sensory block of the upper extremity | within 45 minutes after the block at 5 minutes interval
  Sensation to coldness (ice) will be tested at the median (lateral three and half digits on the palmar side), radial (dorsal side of hand), ulnar (medial one and a half digits), musculocutaneous (lateral side of the forearm), axillary (skin over the lower deltoid) and supra scapular nerve (skin over the scapula) and graded using a verbal rating scale (VRS: 0-100, 100=normal sensation, 0=no sensation). Onset of sensory block for each nerve will be defined as the time that it took to achieve a sensory block score of ≤ 30.
Changes of motor blockade of the upper extremity | within 45 minutes after the block at 5 minutes interval
  Motor blockade will be graded using a 3-points scale revising from previous study: 2 = no block, 1 = paresis and 0 = paralysis. Motor blockade of each individual nerve in the anaesthetized upper extremity will be evaluated by testing for opposition of thumb with the index finger (median nerve), wrist extension (radial nerve), thumb opposition with little finger (ulnar nerve), elbow flexion (musculocutaneous nerve) and abduction of shoulder (axillary nerve). The onset of motor block for each nerve will be defined as motor grading at each nerve ≤ 1. Complete block will be defined as a sensory and motor block score of '0' in all five nerve (median, ulnar, radial, musculocutaneous nerve and axillary) functions and a sensory score of '0' at Suprascapular nerve dermatome.
Readiness for surgery | within 45 minutes after the block at 5 minutes interval
  Overall sensory scores ≤ 30 (VRS: 0-100, 100=normal sensation, 0=no sensation) and motor score ≤ 1 (3-points scale: 2=no block, 1=paresis, 0= paralysis) in all the five nerves tested.

SECONDARY OUTCOMES:
Changes of the Diaphragmatic function | Baseline(before brachial plexus block) and at 30 minutes after block
  Excursion of the right Hemidiaphragm will be measured by ultrasound machine in supine position via the anterior subcostal route. The movement of the diaphragm will be measured in centimetres. The range of diaphragmatic excursion will be recorded from the resting expiratory position to deep inspiration (sigh test) as will be the range of diaphragmatic movement from resting expiratory position when quickly inspiring through the nose (sniff test). The decrease in diaphragmatic excursion will be calculated as the difference (in %) in diaphragmatic excursion measured before and 30 minutes after SeTB. Reduction in diaphragmatic excursion of more than 75%, or no movement, or paradoxical movement will be considered as complete paresis. Reduction in diaphragmatic excursion of both sigh and sniff test between 25% and 75% will be considered as partial paresis and diaphragmatic excursion of less than 25% will be considered as 'no paresis.

CONTACTS AND LOCATIONS:
Overall Officials: Manoj K Karmakar, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Anaesthesia & Intensive Care, Prince of Wales Hospital, Shatin, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No